CLINICAL TRIAL: NCT02185807
Title: Does Video-assisted Informed Consent for Cataract Surgery Improve Patients' Satisfaction
Brief Title: Video-assisted Informed Consent for Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou First People's Hospital (Other)
Responsible Party: Principal Investigator, Yuehong Zhang, Dr., Guangzhou First People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GZFPH-IRB-2013-087
Record Dates: First submitted 2014-07-07; First posted 2014-07-10 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Cataract; Surgery
Keywords: cataract; surgery; consent process; video-assisted
MeSH Terms: conditions — Cataract | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- video-assisted group (Active Comparator): The video assistance patients watch a video in Cantonese or Mandarin explaining the surgery procedure and its risks, benefits and alternatives before discussion with their physicians, and receive face- to face discussion with their physicians as well.
  Interventions: Procedure: video-assisted group
- control group (Placebo Comparator): The control patients receive verbal information and discussion from their physicians.
  Interventions: Procedure: control group

INTERVENTIONS:
Procedure: video-assisted group — The video assistance patients watch a video in Cantonese or Mandarin explaining the surgery procedure and its risks, benefits and alternatives before discussion with their physicians.
  Arms: video-assisted group
Procedure: control group — The control patients receive verbal information and discussion from their physicians.
  Arms: control group

SUMMARY:
The investigators will investigate whether video-assisted informed consent is superior to routine discussion for cataract patients about risks, benefits and alternatives to receiving phacoemulsification cataract extract and intraocular lens implantation, and will determine whether video-assisted informed consent can reduce the work load of physicians.

DETAILED DESCRIPTION:
Patients with age-related cataract who scheduled for elective phacoemulsification cataract extract and intraocular lens implantation surgery and their physicians who on charge of these patients will be enrolled in the study. Patients will be randomized to the video assistance group watched a video in Cantonese or Mandarin explaining the surgery procedure and its risks, benefits and alternatives before discussion with their physicians. The control group will receive traditional verbal information and discussion from their physicians. A questionnaire for patients will be administered to assess the comprehension and satisfaction with the informed consent process before surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients with age-related cataract scheduled for elective phacoemulsification and intraocular lens implantation for the first time in Department of Ophthalmology, Affiliated Hospital of Guangdong Medical College will be recruited in this study. Recruited patients shall own normal intelligence and understanding capability and their best corrected visual acuity more than 0.1 in either eye.

Exclusion Criteria:

Patients who have undergone previously cataract surgery or whose best corrected visual acuity is lower than 0.1 in either eye or patients who complicated with complex other eye diseases such as uveitis and retinal detachment or patients whose language is not cantonese or mandarin will be excluded from this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-07; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
overall patients satisfaction with informed concent | The same day after the surgery

SECONDARY OUTCOMES:
The proportion of patients refusing to sign consent | The same day of surgery
  The proportion of patients who refuse to sign consent for the surgery
A 10-question cataract surgery knowledge measure | The same day after the surgery
  A written examination (0% to 100%) on patient understanding of the risks, benefits, and alternatives of cataract surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yuehong Zhang, MD, PhD, Principal Investigator — Guangzhou First People's Hospital; Min Lu, MD, Principal Investigator — Sanshui District People's Hospital of Foshan
Locations (2):
- China (2):
  - Sanshui District People's Hospital of Foshan;Guangzhou First Peoples' Hospital, Affiliated Hospital of Guangzhou Medical University, Foshan, Guangdong
  - Guangzhou First Municipal People's Hospital, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided